CLINICAL TRIAL: NCT04101643
Title: PCSK9 Inhibitor Treatment for Patients With Hereditary Spastic Paraplegia Type 5
Brief Title: PCSK9 Inhibitor Treatment for Patients With SPG5
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Wan-Jin Chen, Neurology department, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MRCTA, ECFAHofFMU[2019]209
Record Dates: First submitted 2019-09-22; First posted 2019-09-24 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Hereditary Spastic Paraplegia Type 5
MeSH Terms: interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evolocumab group (Experimental): Eligible patients receive subcutaneous injections of evolocumab 420 mg
  Interventions: Drug: evolocumab

INTERVENTIONS:
Drug: evolocumab — Eligible patients receive subcutaneous injections of evolocumab 420 mg

SUMMARY:
Spastic paraplegia type 5 (SPG5) is a rare subtype of hereditary spastic paraplegia, a highly heterogeneous group of neurodegenerative disorders defined by progressive neurodegeneration of the corticospinal tract motor neurons. SPG5 is caused by recessive mutations in the gene CYP7B1 encoding oxysterol-7a-hydroxylase. This enzyme is involved in the degradation of cholesterol into primary bile acids. CYP7B1 deficiency has been shown to lead to accumulation of neurotoxic oxysterols. Oxysterols were found to impair metabolic activity and viability of human cortical neurons at concentrations found in SPG5 patients, indicating that elevated levels of oxysterols might be key pathogenic factors in SPG5. Monoclonal antibodies that inhibit proprotein convertase subtilisin-kexin type 9 (PCSK9) have emerged as a new class of drugs that effectively lower cholesterol levels. Evolocumab, a member of this class, is a fully human monoclonal antibody that reduces LDL cholesterol levels by approximately 60%. We thus performed this interventional trial with Evolocumab 420 mg for SPG5 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-80 years
* Probands with clinically manifest hereditary spastic paraplegia
* Genetically confirmed diagnosis of SPG5

Exclusion Criteria:

* Comprised treatment with statins 3 months prior to enrolment
* Contraindications to PCSK9 inhibitor therapy
* Pregnancy was excluded in women of childbearing age

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-29 (Actual); Primary Completion 2023-01-03 (Estimated); Study Completion 2023-01-03 (Estimated)

PRIMARY OUTCOMES:
The change of 27-hydroxycholesterol (27-OHC) | up to 4 weeks
  Cholesterol is initially side chain oxidized and the resulting 27-hydroxycholesterol (27-OHC) are 7a-hydroxylated

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Jin Chen, Principal Investigator — First Affiliated Hospital Fujian Medical University
Locations (1):
- Department of Neurology , First Affiliated Hospital Fujian Medical University, Fuzhou, China